CLINICAL TRIAL: NCT00573300
Title: Disturbances of Kynurenine Pathway of Trytophan Metabolism in Schizophrenia: A Quantitative RT-PCR Study
Brief Title: Disturbances of Kynurenine Pathway of Trytophan Metabolism in Schizophrenia: A Quantitative Reverse Transcription Polymerase Chain Reaction (RT-PCR) Study
Status: Completed | Type: Observational
Sponsor: North Suffolk Mental Health Association (Other)
Responsible Party: Oliver Freudenreich, MD, Massachusetts General Hospital
Other Study IDs: CORRC#10-2005
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2009-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Immune System; Kynurenate; tryptophan metabolism; NMDA receptor; indolamine 2,3-deoxygenase (IDO)
MeSH Terms: conditions — Schizophrenia | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Schizophrenia: Schizophrenia Patients
  Interventions: Procedure: Phlebotomy
- Healthy Controls: Healthy Controls
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Single blood draw

SUMMARY:
In this pilot study, the investigators propose to characterize the pattern of activation of the kynurenine pathway of tryptophan metabolism in peripheral macrophages of patients with schizophrenia. To do this, the investigators will measure the gene expression of several major enzymes in this pathway in macrophages, including the key enzyme involved in tryptophan to kynurenine metabolism, IDO, by means of quantitative reverse-transcription polymerase chain reaction (RT-PCR). The focus on enzyme mRNA expression as opposed to serum or cerebrospinal fluid levels of metabolites provides a possibly more sensitive characterization of the activation of this metabolic pathway.

DETAILED DESCRIPTION:
In this pilot study, we propose to characterize the pattern of activation of the kynurenine pathway of tryptophan metabolism in peripheral macrophages of patients with schizophrenia. To do this, we will measure the gene expression of several major enzymes in this pathway in macrophages, including the key enzyme involved in tryptophan to kynurenine metabolism, IDO, by means of quantitative reverse-transcription polymerase chain reaction (RT-PCR). The focus on enzyme mRNA expression as opposed to serum or cerebrospinal fluid levels of metabolites provides a possibly more sensitive characterization of the activation of this metabolic pathway.

Primary hypotheses: We hypothesize that patients with schizophrenia will differ in their expression of macrophage IDO mRNA, reflecting activation of this pathway compared to normals. We further hypothesize that patients with deficit syndrome will have higher degrees of enzyme activation.

Secondary hypotheses: Serum tryptophan levels will be lower in patients with schizophrenia compared to controls, and they will correlate with measures of dysphoria. Serum kynurenine levels will be elevated in patients with schizophrenia, particularly in deficit syndrome patients. mRNA expression levels of enzymes downstream from IDO will differ between patients and controls. Measures of immune activation will be influenced by medical disease burden (medical comorbidities).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Schizophrenia, any subtype or schizoaffective disorder
2. Ages 18-65 years
3. Males or females
4. English speaking with ability to complete symptom ratings
5. Ability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Schizophrenia patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Freudenreich, M.D., Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States